CLINICAL TRIAL: NCT05610800
Title: A Randomized Controlled Trial of Exenatide as an Adjunct to Nicotine Patch for Smoking Cessation and Prevention of Post-Cessation Weight Gain
Brief Title: Exenatide for Smoking Cessation and Prevention of Weight Gain
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Luba Yammine, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-21-0639
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation; Weight Gain
Keywords: Smoking; Cigarettes; Nicotine; Cigarette Smoking; Weight Gain Prevention; Post-cessation Weight Gain
MeSH Terms: conditions — Smoking Cessation; Weight Gain; Smoking; Cigarette Smoking | interventions — Injections; Exenatide; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exenatide, NRT, and Smoking Cessation Counseling (Active Comparator): Participants will receive once weekly exenatide injections, daily nicotine patches (NRT), and once weekly individual smoking cessation counseling sessions.
  Interventions: Drug: Exenatide 2 milligram (mg) Injection; Drug: Nicotine patch; Behavioral: Smoking Cessation Counseling
- Placebo, NRT, and Smoking Cessation Counseling (Placebo Comparator): Participants will receive once weekly saline injections, daily nicotine patches (NRT), and once weekly individual smoking cessation counseling sessions.
  Interventions: Drug: Placebo; Drug: Nicotine patch; Behavioral: Smoking Cessation Counseling

INTERVENTIONS:
Drug: Exenatide 2 milligram (mg) Injection — Exenatide will be purchased commercially as Bydureon for subcutaneous (SC) injection and administered at a dose of 2 mg once a week for a total of 14 weeks. Each single-dose, dual-chamber pen contains 0.65 mg of diluent and 2 mg of exenatide, which remains isolated until mixed.
  Other Names: Bydureon
  Arms: Exenatide, NRT, and Smoking Cessation Counseling
Drug: Placebo — Sterile saline (0.9%) will serve as the placebo for exenatide. The placebo will be administered 2 mg subcutaneously using insulin syringes.
  Arms: Placebo, NRT, and Smoking Cessation Counseling
Drug: Nicotine patch — Nicotine patches will be purchased commercially and dispensed during clinic visits for one week of use.
  Participants who smoke >10 cigarettes/day will receive 21 mg patches for the first 12 weeks, 14 mg patches for week 13, and 7 mg patches for week 14.
  Participants who smoke 5-10 cigarettes per day will receive 14 mg patches for the first 12 weeks and 7 mg patches for weeks 13 and 14.
Behavioral: Smoking Cessation Counseling — Participants will receive brief individual behavioral smoking cessation counseling that consist of weekly in-person sessions and 2 brief (10-15 min) supportive phone calls (once pre-quit and again 3-days post-quit), spanning the 14-week active treatment phase. Counseling will be provided by master's level clinicians who will receive at least 8 hours of initial training.

SUMMARY:
The purpose of this study is to determine if exenatide improves end-of-treatment smoking abstinence rates and to determine if exenatide mitigates post-cessation weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to sign and date an informed consent form, willing to comply with all study procedures, and be available for the duration of the study
* Male or female, 18-75 years of age
* Have been smoking ≥5 cigarettes per day for at least 1 year and provide positive cotinine test
* Desire to quit smoking (defined as "intend to quit within one month")
* Have HbA1C levels between 5.7 and 6.4% and/or a body mass index of ≥25 kg/m2
* Have vital signs as follows: resting pulse between 50 and 95 bpm, BP between 90-150 mmHg systolic and 45-95 mmHg diastolic
* Have hematology and chemistry laboratory tests that are within reference limits (±10%), with the following exception: pancreatic tests (lipase and amylase) must be within normal limits
* Agree (if the subject is female and of child-bearing potential) to use at least one of the following methods of birth control from time of the first administration of the study medication to at least 7 days post the last dose of the study medication, unless the partner is surgically sterile (underwent vasectomy): oral contraceptives, contraceptive sponge, patch, double barrier (diaphragm/spermicidal or condom/spermicidal), intrauterine contraceptive system, etonogestrel implant, medroxyprogesterone acetate contraceptive injection, hormonal vaginal contraceptive ring, or complete abstinence from sexual intercourse.
* Women of child-bearing potential must provide negative urine pregnancy tests prior to randomization
* Have a medical history and a brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the Study Physician and the PI.

Exclusion Criteria:

* Psychoactive substance abuse or dependence (excluding nicotine dependence) within the past 3 months (existing diagnosis or as determined by the structured interview)
* Currently using chewing tobacco, snuff, snus or electronic cigarettes
* Currently enrolled in a smoking cessation program/research study or using pharmacotherapy for smoking cessation (NRT, varenicline, or bupropion)
* Currently enrolled in a behavioral weight management plan/research study, or taking medication used for weight management (i.e., orlistat, lorcaserin,*naltrexone-bupropion, liraglutide, phentermine, benzhetamine, diethylpropion, phendimetrazine), or medication known to impact weight (i.e., corticosteroids) *Note: Withdrawn from the market in Feb 2020, but some patients may still be taking it
* Currently using oral or injectable glucose lowering medications
* Urine drug test positive, before randomization, for any of the following substances: benzodiazepines, cocaine, opioids,*amphetamines, methamphetamine, buprenorphine, barbiturates, 3,4-methylenedioxy-methamphetamine (MDMA), and/or THC. *Note: If positive for opioids or oxycodone but recent opioid use for acute pain is reported by the study candidate, then the candidate can be included at the discretion of the Primary Investigator and/or Study Physician
* Psychotic or bipolar disorder, or mood disorder with psychotic features, or eating disorder (existing diagnosis or as determined by the structured interview)
* Moderate to high risk for suicidality (as determined by the structured interview)
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2)
* Type 1 or type 2 diabetes mellitus (previously diagnosed or indicated by HbA1C level of ≥6.5%)
* Severe cardiovascular disease (history of myocardial infarction, life-threatening arrhythmia, or worsening angina pectoris)
* Severe gastrointestinal disease (i.e., severe gastroparesis)
* Previous history of pancreatitis or risk of pancreatitis
* Creatinine clearance <45 mL/min or end stage renal disease (ESRD)
* Previous medically adverse reaction to the study medications or nicotine
* Women who are currently pregnant, or plan to become pregnant, or lactating, or of childbearing potential and are not using medically accepted forms of contraception. Medically accepted forms of contraception are specified in the inclusion criterion 8.
* Current, anticipated, or pending enrollment in another research study over the next 6 months that could potentially affect subject safety and/or the study data/design as determined by the PI and/or Study Physician
* Unable to communicate (read, write, and speak) fluently in English
* Have any illness or condition which in the opinion of the PI and/or the Study Physician would preclude safe and/or successful completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with 4-week continuous abstinence at 12 weeks post-target quit day as assessed by self-report timeline followback (TLFB) and verified by breath carbon monoxide (CO) level | Week 15
  Abstinence is defined as no smoking, not even a puff, as reported on TLFB between weeks 11 through 14 and biochemically verified (CO ≤ 5 ppm) at each visit.
Weight change in kilograms at 12 weeks post-target quit day | Baseline, Week 15

SECONDARY OUTCOMES:
Percentage of participants with 4-week continuous abstinence at 24 weeks post-target quit day as assessed by self-report timeline followback (TLFB) and verified by breath carbon monoxide (CO) level | Week 26
  Abstinence is defined as no smoking, not even a puff, as reported on TLFB between weeks 22 through 25 and biochemically verified (CO ≤ 5 ppm) at Week 26.
Weight change in kilograms at 24 weeks post-target quit day | Baseline, Week 26
Change in amplitude of the late positive potential evoked by visual stimuli | Week 1, Week 3

CONTACTS AND LOCATIONS:
Overall Officials: Luba Yammine, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yammine L, Verrico CD, Versace F, Webber HE, Suchting R, Weaver MF, Kosten TR, Alibhai H, Cinciripini PM, Lane SD, Schmitz JM. Exenatide as an adjunct to nicotine patch for smoking cessation and prevention of postcessation weight gain among treatment-seeking smokers with pre-diabetes and/or overweight: study protocol for a randomised, placebo-controlled clinical trial. BMJ Open. 2023 Jun 14;13(6):e072707. doi: 10.1136/bmjopen-2023-072707. PMID 37316311